CLINICAL TRIAL: NCT07073417
Title: A Multicenter, Randomized, Open-label, Treatment Switching Phase II Study to Evaluate the Efficacy and Safety of XW003 Injection and Semaglutide Injection in Chinese Adults With Obesity
Brief Title: A Study to Compare XW003 Injection and Semaglutide Injection in Chinese Adults With Obesity (SLIMMER-UP-SWITCH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCW0502-1122
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Weight Management
Keywords: Weight management; obesity; XW003; glucagon-like peptide-1 (GLP-1); ecnoglutide; semaglutide
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XW003 (Experimental): once weekly
  Interventions: Drug: XW003 injection
- semaglutide (Active Comparator): once weekly
  Interventions: Drug: semaglutide injection

INTERVENTIONS:
Drug: XW003 injection — Subcutaneous injection
  Other Names: ecnoglutide
  Arms: XW003
Drug: semaglutide injection — Subcutaneous injection
  Arms: semaglutide

SUMMARY:
The aim of the study is to compare the efficacy and safety of XW003 injection versus semaglutide injection in Chinese adults with obesity

DETAILED DESCRIPTION:
In this Phase II study, eligible participants will be randomized into one of the two cohorts in a 1:1 ratio to receive once-weekly subcutaneous XW003 injection or semaglutide injection, including a dose-escalation period, a core treatment period and a treatment extension period, for up to 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥30 kg/m2 at screening, waist circumference ≥90 cm for men and ≥85 cm for women.
* Weight change of less than 5% within 3 months prior to screening (self-reported).

Exclusion Criteria:

* Diagnosis of obesity due to endocrine disorders or a single gene mutation, including but not limited to hypothalamic obesity, pituitary obesity, Cushing's syndrome, hypothyroidic obesity (except for those with normal thyroid function at screening and expected to remain unchanged throughout the trial period after at least 3 months of thyroid hormone replacement therapy), insulinoma, acromegaly.
* History of bariatric surgery or planning to undergo bariatric surgery or use other weight-loss drugs or devices during the trial (except acupuncture for weight loss, liposuction, or abdominal fat removal for more than one year before screening; Except the removal or expulsion of the airbag in the stomach for more than 1 year before screening.
* Diagnosis with any type of diabetes (except gestational diabetes).
* Have used any weight-loss drugs, hypoglycemic drugs, or drugs that may cause significant weight gain within 3 months prior to screening.
* History of acute or chronic pancreatitis or pancreatic injury, history of symptomatic gallbladder disease (except cholecystectomy).
* History of clinically significant gastric emptying abnormalities, such as gastroparesis or gastric outlet obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight relative to baseline | week 48

SECONDARY OUTCOMES:
Proportions of participants with weight loss ≥5% from baseline | week 48
Proportions of participants with weight loss ≥10% from baseline | week 48
Proportions of participants with weight loss ≥15% from baseline | week 48
The change in waist circumference relative to the baseline | week 48
Changes in body mass index (BMI) relative to baseline | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Dr, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China